CLINICAL TRIAL: NCT01512017
Title: A Clinical Study to Evaluate the Safety and Efficacy on Veloderm (a Crystalline Cellulose Simple Occlusive Dressing) for the Split-thickness Skin Graft Donor Sites in Burn and Plastic Surgery
Brief Title: Clinical Study on Veloderm for the Treatment of Split-thickness Skin Graft Donor Sites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Ruijin Hospital (Other); Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZHAOKE-VL2010
Record Dates: First submitted 2010-09-14; First posted 2012-01-19 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Split-thickness Skin Graft Donor Sites
Keywords: skin lesions or defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Veloderm (Active Comparator)
  Interventions: Device: Crystalline cellulose simple occlusive dressing
- Vaseline (Placebo Comparator)
  Interventions: Device: Vaseline

INTERVENTIONS:
Device: Crystalline cellulose simple occlusive dressing — A natural biological film of vegetable origin. It is classified as skin semi occlusive dressing, as a temporary skin substitute in case of skin lesions or loss.
  Other Names: Veloderm
  Arms: Veloderm
Device: Vaseline — External use
  Arms: Vaseline

SUMMARY:
This study is a multi-center, randomized, open and paralleled positive control study for evaluating the safety and efficacy of Veloderm in treatment of split-thickness skin graft donor sites. The result implies that Veloerm can do it better than Vaseline gauze in accelerating and promoting wound healing of skin graft donor sites. The present study have indicated that high permeability of Veloderm dressing to oxygen and water vapor.

DETAILED DESCRIPTION:
The rational oxygen permeability of Veloderm dressing also provides a good environment for wound healing. Therefore, it can be as a temporary skin substitute in the case of missing epidermis to play a role, in order to provide an ideal environment for wound epithelialization. As regards safety, 1 adverse reaction occured in test group. It shows effusion under the dressing mild inflammatory infiltration on the wound edge. After the dressing was changed and the effusion was drained, the patient was relieved. As Veloderm dressing itself has no direct anti-inflammatory effects, clinical application as appropriate can plus other anti-infective drugs in accordance with patient conditions. In conclusion, Veloderm is a safe and effective dressing to accelerate the healing of donor sites in burn and plastic surgery. Veloderm can be used as a temporary skin substitute in case of damage of skin or loss of superficial epidermal (such as burns, wounds, abrasions, ulcers, sores and auto-graft donor areas).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Male or female patients
* Skin lesions or losses by burns, plastic surgery, sores, abrasions, donor graft areas and after debridement of chronic wounds
* The area of skin loss or burn surface is less than 50% of total area of body surface
* Subject undergoing first skin harvest 0.25-0.35mm and donor site having a surface area>100cm2
* Subject who is willing to participate in the trial and to sign the informed consent form.

Exclusion Criteria:

* Area of skin loss or burn surface is larger than 50% of total area of body surface
* Electrical burns or chemical burns
* Burns complicated by combined injury
* Test wound needs drugs that may affect wound healing
* Subject who has a known hypersensitivity to hemycellulose
* Contraindication to the use of semi occlusive dressing
* Pregnant or lactating subject
* Any severe disease which in the Investigator's judgement might interfere with study evaluations or threaten patient's safety
* Subject who has chronic renal disease or renal inadequacy, or serum creatinine is more than twice the upper limit of normal
* Subject who has a definite liver disease, TBil or AST, ALT is more than twice the upper limit of normal
* Subject with active hemorrhoea or shock or visceral injury; Subject who has participated in this clinical study or other clinical studies within 3 months
* Subject with mental impairment limiting the ability to comply with study requirements; Subject undergone chronic treatment with immunosuppressants, antineoplastic drugs and corticosteroids for a long time
* Subject who has not signed the informed consent form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Response Criteria | 3 months
  To observate the efficacy measurements, vital signs, laboratory examinations and adverse events

SECONDARY OUTCOMES:
Evaluation criteria | 6 months
  To evaluate the time to complete epithilization, effectiveness, presence of exudates, presence of prei-lesional erythema, pain intensity and laboratory examination